CLINICAL TRIAL: NCT03528616
Title: Management of Supraventricular Tachycardia of Children Admitted to Assiut University Children Hospital(Clinical Audit)
Brief Title: Management of Supraventricular Tachycardia of Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Hussien, principal investigator, Assiut University
Other Study IDs: SVT
Record Dates: First submitted 2018-04-20; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Adenosine; Amiodarone; Propranolol; Digoxin; Procainamide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: adenosine,Propranolol,flecainide, amiodarone, propranolol, digoxin and procainamide. — drugs used for treatment of supraventricular tachycardia

SUMMARY:
• Supraventricular tachycardia (SVT) is defined as an abnormally rapid heart rhythm originating above the ventricles. It usually has narrow complex tachycardia but this is not always the case. Conventionally, atrial flutter and fibrillation are excluded from this group.ventricular tachycardia is the most common rhythm disturbance seen in children.(2) Most general practitioners will deal with a case at some point. While in most cases ventricular tachycardia can be considered a benign rhythm disorder, special consideration needs to be given to infants, athletes and patients with Wolff-Parkinson-White syndrome.

DETAILED DESCRIPTION:
Epidemiology Incidence of Supraventricular tachycardia is estimated to occur in 1 in 250 otherwise healthy children. About 50% of children with Supraventricular tachycardia present with the first episode in the first year of life.

After infancy there is another surge in incidence in early childhood (6-9 years) and then in adolescence.In more than 90% of infants spontaneous resolution occurs by 1 year of age but up to a third have a subsequent recurrence of Supraventricular tachycardia at a mean age of 8 years. Spontaneous resolution is uncommon (15%) in those presenting after 1 year of age.

Most children with Supraventricular tachycardia have a structurally normal heart but the prevalence of congenital heart disease in patients with Supraventricular tachycardia is substantially higher than that of the general population (9-32%).

Clinical presentation Clinical presentation depends on the age of the child and the duration of Supraventricular tachycardia.

In infants the heart rate is usually about 220 to 320 bpm and symptoms are usually nonspecific, including poor feeding, irritability, vomiting and dusky episodes. If the symptoms are unrecognised for hours or days the infant may present with heart failure or shock.In older children the heart rate is between 160 to 280 bpm and the usual presenting symptoms are palpitations, chest pain and shortness of breath. Often light-headedness and dizziness can occur; however, syncope is rare.

The frequency and duration of episodes can vary hugely, with episodes lasting a few minutes to several hours and occurring once a year to several times a day.

Physical examination is normal apart from the infant presenting in heart failure and shock.

Investigations

Diagnosis is confirmed by making an ECG recording during symptoms. Options available for this are:

Holter (24-hour ambulatory ECG) monitoring in children having daily symptoms. Cardiac event recorders in those who have brief infrequent symptoms. ECG in the emergency department (ED) in those with infrequent but prolonged symptoms allowing them to travel to ED in the event of symptoms.

ECG done during episodes is diagnostic and shows:

Tachycardia with narrow QRS complexes. P waves may not be visible. If visible, they exhibit retrograde conduction with inverted P waves.A baseline echocardiography to confirm the presence of a structurally normal heart and to ensure that,heart function is normal,is recommended.

Acute management of Supraventricular tachycardia Acute management of Supraventricular tachycardia is primarily based on use of vagal manoeuvres and/or adenosine. Sometimes other medications and occasionally direct current (DC) shock are needed.

Advanced Paediatric Life Support guidelines recommend the following approach:

Assess airway, breathing and circulation (ABC) in any child or infant presenting with Supraventricular tachycardia. Try vagal stimulation while continuing ECG monitoring. The techniques that can be used include:

Elicit the 'diving reflex' by applying a rubber glove filled with iced water on the face or wrapping the infant in a towel and immersing the face in iced water for five seconds.

One-sided carotid massage. Valsalva manoeuvre in older children. Give IV adenosine if vagal manoeuvres are unsuccessful. Start with a bolus dose of 100 micrograms/kg intravenously. If this does not work, increasing doses (200 micrograms/kg and then 300 micrograms/kg) can be given after two minutes. The maximum single dose that is given is 500 micrograms/kg (300 micrograms/kg in infants less than 1 month of age), up to a maximum of 12 mg.

In a hemodynamically stable child not responding to adenosine, alternative medications should be used based on advice by a paediatric cardiologist. The options available include flecainide, amiodarone, propranolol, digoxin and procainamide.

verapamil has been associated with irreversible hypotension and asystole in infants and should not be used in this age group.

Wide complex Supraventricular tachycardia(i.e Supraventricular tachycardia with aberrant conduction) is uncommon in infants and children.

In an infant or child with Supraventricular tachycardia and in shock the best treatment option is synchronised DC cardioversion starting at a dose of 1 joule/kg and increasing to 2 joules/kg if necessary.

Long-term management Long-term management is dependent on a number of factors, including the age of patient, duration and frequency of episodes and presence of ventricular dysfunction. Management is carried out under the supervision of a pediatric cardiologist.In children with infrequent, mild and self-limiting episodes, usually no treatment is needed.In children in whom the episodes are frequent, prolonged, difficult to terminate or interfering with sports participation, treatment is indicated. Treatment options include medications or transcatheter ablation.

1. Medical treatment The purpose of using anti-arrhythmic drugs is to slow conduction, preferentially within one limb of the re-entrant circuit and therefore terminate the tachycardia.

   Treatment options include digoxin, beta-blockers, calcium-channel blockers and the sodium-channel blocker, flecainide.

   While there is significant variation in practice, the majority of European centers use flecainide or atenolol as the first choice of drug for the prevention of recurrent Supraventricular tachycardia.

   There is little difference in the efficacy of various medications and a randomised controlled trial comparing digoxin and propranolol found no difference in recurrence of Supraventricular tachycardia in the two groups.

   While any of the anti-arrhythmics can be used to initiate treatment.
2. Ablation treatment Management of Supraventricular tachycardia has been revolutionised with the development of transcatheter ablation which is now considered standard treatment for older children and adolescents.

Radiofrequency (RF) is the preferred energy source for paediatric arrhythmias and catheter ablation is only chosen if two or more anti-arrhythmic drugs have failed.

An alternative to RF is cryoablation, which is safer and minimises the risk of heart block during ablation. However, it is associated with a higher Supraventricular tachycardia recurrence rate and therefore most centers use cryoablation in cases where RF ablation is considered a higher risk.

Sports participation and general advice Patients and parents should be reassured that Supraventricular tachycardia is typically not life-threatening but can be life-altering.

Parents and patients should be taught age-appropriate vagal manoeuvres and indications for requesting assistance from emergency services. These include:

Prolonged symptoms. Episode not terminated by vagal manoeuvres. Syncope.

Routine school physical activities including recreational sports participation are allowed.Much more caution needs to be exercised in those participating in competitive athletics and high-speed or contact sports. Guidelines issued by the American Heart Association recommend the following:

Asymptomatic athletes with structurally normal hearts and exercise-induced Supraventricular tachycardia prevented by medical treatment can participate in all competitive sport.

Athletes who have had successful transcatheter ablation and are asymptomatic with no inducible arrhythmia can return to full competition.

Fetal supraventricular tachycardia It accounts for 60%-80% of fetal tachyarrhythmias, with prevalence ranging from 1 in 1,000 to 1 in 25,000 pregnancies.

Clinical presentation is variable. Intermittent Supraventricular tachycardia may have no hemodynamic effect, while persistent Supraventricular tachycardia may result in fetal hydrops due to high-output cardiac failure.

Risk of developing hydrops is related to the age of the fetus (the younger is more susceptible) and duration of Supraventricular tachycardia.

Diagnosis is made by fetal echocardiography using M mode and Doppler. Treatment is transplacental therapy with anti-arrhythmics such as digoxin and flecainide.

Prognosis:

In the absence of structural heart disease or cardiomyopathy, the prognosis of Supraventricular tachycardia is excellent.

ELIGIBILITY:
Inclusion Criteria:

* Cases of SVT who will be admitted to Assiut University Children hospital during the period between May,2018 to May,2019.

Exclusion Criteria:

* newborns up to one month age

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: prospective observational study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate management of SVT in the cardiology unit of Assiut University Children Hospital according to international guidelines by using pharmacological and non pharmacological treatments. | one year
  Descriptive sheet of the study checklist that will be asked about in all cases: Clinical examination and ECG at presentation,Physical maneuvers(vagal stimulation),Drug therapy including:adenosine and other antiarrythmic drugs as Flecainide,propranolol,amiodarone,digoxin and verapamil.
  Appropriate dose of drugs,Putting on monitor ECG during treatment,Synchronized DC cardioversion in hemodynamically unstable cases.
  Yes ,No ,℅ of the folowing, Clinical examination and ECG at presentation Vagal manoeuvers,diving reflex,One side carotid massage,Valsalva manoeuvre Drug therapy Adenosine only,Flecainide only,Propranolol and Amiodarone,Amiodarone only Digoxin only,Digoxin then Amiodarone, Verapamil Maintain ECG monitoring,Synchronized DC cardioversion. These data will be collected and revised to show how would doctors in the cardiology unit of Assiut University Children Hospital manage SVT according to the international guinternational guidelines.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sawhney V, Corden B, Abdul-Mukith K, Harris T, Schilling RJ. Are patients admitted to emergency departments with regular supraventricular tachycardia (SVT) treated appropriately? Clin Med (Lond). 2013 Apr;13(2):146-8. doi: 10.7861/clinmedicine.13-2-146. PMID 23681861